CLINICAL TRIAL: NCT06361745
Title: Early Clinical Study of UTAA09 Injection in the Treatment of Relapsed/Refractory
Brief Title: Early Clinical Study of UTAA09 Injection in the Treatment of Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-005-6
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus; Idiopathic Inflammatory Myopathies; Systemic Sclerosis; IgG4 Related Disease; Primary Sjögren Syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis; Scleroderma, Systemic; Immunoglobulin G4-Related Disease

STUDY DESIGN:
Intervention Model Description: UTAA09 injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T cell injection targeting CD19 chimeric antigen receptor (Experimental): Intravenous administration, 1 bag each time (depending on individual differences), dose: 1×108-1×109 CD19-CAR-gdT (UTAA09 injection), the investigator can decide whether to reduce or increase the dose and whether multiple infusions are required according to the condition of the subject
  Interventions: Biological: T cell injection targeting CD19 chimeric antigen receptor

INTERVENTIONS:
Biological: T cell injection targeting CD19 chimeric antigen receptor — Intravenous administration, 1 bag each time (depending on individual differences), dose: 1×108-1×109 CD19-CAR-gdT (UTAA09 injection), the investigator can decide whether to reduce or increase the dose and whether multiple infusions are required according to the condition of the subject.

SUMMARY:
Main purpose:

To evaluate the safety of UTAA09 injection in the treatment of relapsed/refractory (R/R) autoimmune disease (AID).

Secondary purpose:

To evaluate the pharmacokinetic (PK) profile of UTAA09 injection in patients with R/R AID.

To evaluate the pharmacodynamic (PD) characteristics of UTAA09 injection in patients with R/R AID.

To evaluate the initial efficacy of UTAA09 injection in the treatment of R/R AID subjects.

To evaluate the immunogenicity of UTAA09 injection in R/R AID subjects.

DETAILED DESCRIPTION:
This clinical trial was designed as a single-arm, open-label, single-center, investigator-initiated early-stage clinical study to evaluate the safety of UTAA09 injection in patients with relapsed/refractory AID. After signing the informed consent letter, qualified subjects were screened for infusion of UTAA09 injection, and their blood was collected before and after infusion for pharmacokinetics, pharmacodynamics, immunogenicity, safety and other evaluation. In addition to the baseline period, the therapeutic efficacy was evaluated at the frequency of 14d, 28d, 2m, 4m, 6m, 8m, 10m, 12m, 15m, 18m, 21m, 24m after cell transfusion until disease progression (PD), new anti-disease therapy, death, intolerable toxicity, investigator decision, or subject's voluntary withdrawal. Whichever comes first.

ELIGIBILITY:
inclusion criteria (2) Expected survival time ≥3 months; (3) Subjects with recurrent/refractory autoimmune diseases who have failed standard treatment or lack effective treatment, Including but not limited to systemic lupus erythematosus, idiopathic inflammatory myopathy, systemic sclerosis, IGG4-associated diseases, primary Sjogren's syndrome, rheumatoid arthritis, connective tissue disease-associated interstitial lung disease, immune thrombocytopenia, primary biliary cholangitis, etc.

(3) Histological evidence of non-suppurative destructive cholangitis and small bile duct destruction.

(4) Liver and kidney function, cardiopulmonary function meet the following requirements:

* Creatinine ≤1.5×ULN; (2) Electrocardiogram showed no clinically significant abnormal bands;

  * Blood oxygen saturation >91% in non-oxygen state;

    * Total bilirubin ≤2×ULN; ALT and AST≤2.5 x ULN; ALT and AST abnormalities due to disease, such as liver infiltration or bile duct obstruction, were determined to be less than 5×ULN. If Gilbert syndrome is diagnosed, the total bilirubin index can be relaxed to ≤3.0×ULN and the direct bilirubin ≤1.5×ULN.

      (5) no serious mental disorders; (6) Can understand this test and have signed the informed consent.

Exclusion criteria:

1. Malignant tumors other than R/R AID disease in the 5 years prior to screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery;
2. Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal reference value range; Hepatitis C virus (HCV) Antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; Human immunodeficiency virus (HIV) Antibody positive; Syphilis positive;
3. Serious heart disease, including but not limited to unstable angina, myocardial infarction or bypass or stent surgery (within 6 months prior to screening), congestive heart failure (NYHA classification ≥III), and severe arrhythmia;
4. Systemic diseases that are deemed unstable by researchers: including but not limited to severe liver, kidney, or metabolic diseases that require drug treatment;
5. Active or uncontrollable infections (except mild genitourinary and upper respiratory tract infections) that require systemic treatment within 7 days prior to administration;
6. Pregnant or lactating women, and female subjects who plan pregnancy within 2 years after cell transfusion or male subjects whose partners plan pregnancy within 2 years after cell transfusion;
7. Patients who received CAR-T therapy or other gene-modified cell therapy before screening;
8. Participated in other clinical studies 1 month before screening;
9. Evidence of central nervous system invasion during subject screening;
10. Mental patients with depression or suicidal thoughts;
11. Those who received live vaccine within 28 days prior to screening;
12. Situations considered unsuitable for inclusion by other researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
AE | 3 months after cell reinfusion or disease progression/recurrence or start of new anti-disease therapy (whichever occurs first)
  Type, frequency, and severity of adverse events (AEs) and laboratory abnormalities according to the Common Adverse Event Evaluation Standard NCI CTCAE version 5.0

SECONDARY OUTCOMES:
Cmax | 3 months after cell reinfusion or disease progression/recurrence or start of new anti-disease therapy (whichever occurs first)
  The maximum amplified concentration (Cmax) of UTAA09 injection in peripheral blood after administration, the time to reach the maximum concentration (Tmax), and the area under the curve AUC0-28d at 28 days and the area under the curve AUC0-90d at 90 days
CD19-positive cells | 3 months after cell reinfusion or disease progression/recurrence or start of new anti-disease therapy (whichever occurs first)
  The content of CD19-positive cells in peripheral blood after UTAA09 injection administration: the proportion and absolute value of CD19-positive cells in peripheral blood at each time point; Concentration levels of CAR-T-associated serum cytokines.
Disease remission/response/improvement rates | 3 months after cell reinfusion or disease progression/recurrence or start of new anti-disease therapy (whichever occurs first)
  Disease remission/response/improvement rates at 28 days, 2 months, and 3 months after administration.
anti-CAR antibody | 3 months after cell reinfusion or disease progression/recurrence or start of new anti-disease therapy (whichever occurs first)
  The positive rate of human anti-CAR antibody at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: songlou yin, master, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- PersonGen.Anke Cellular Therapeutice Co., Ltd, Hefei, China

IPD SHARING:
Plan to Share IPD: No